CLINICAL TRIAL: NCT06876649
Title: A Master Protocol to Evaluate the Long-Term Safety of Pirtobrutinib
Brief Title: A Master Protocol to Evaluate the Long-Term Safety of (LY3527727) Pirtobrutinib
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 27202; 2024-517760-29-00 (EU CTIS Number); J2N-MC-JZNY (Other: Eli Lilly and Company); J2N-MC-JZ01 (Other: Eli Lilly and Company); J2N-MC-JZ02 (Other: Eli Lilly and Company); J2N-MC-JZ03 (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-03-06; First posted 2025-03-14 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Chronic Lymphocytic Leukemia; Non-Hodgkin Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Non-Hodgkin | interventions — pirtobrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- JZ01 Pirtobrutinib (Experimental): Participants receive pirtobrutinib as defined in the originator study (LOXO-BTK-18001/J2N-OX-JZNA).
  Pirtobrutinib administered orally.
  Interventions: Drug: Pirtobrutinib

INTERVENTIONS:
Drug: Pirtobrutinib — Administered orally.
  Other Names: LOXO-305; LY3527727

SUMMARY:
The master protocol study J2N-MC-JZNY provides a framework to enable the evaluation of the long-term safety and efficacy of pirtobrutinib after completion of clinical studies evaluating pirtobrutinib. The clinical studies that will feed into this master protocol are referred to as originator studies. The master protocol will govern individual study-specific appendices (ISAs) that will represent participants from the individual, completed originator studies. These participants will have the opportunity to enter this study and continue to receive treatment or continue follow-up visits. Overall, the master protocol and the individual ISAs, when combined, define the investigations for this study.

ELIGIBILITY:
Inclusion Criteria:

* Are participating in an eligible Lilly sponsored clinical study evaluating pirtobrutinib.

Exclusion Criteria:

Exclusion criteria are defined in each ISA.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 787 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2030-05 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with a Grade ≥3 treatment-emergent AEs | Time from the Date of the First Dose of Study Intervention (Study Day 1) through 30 Days (+ 7-day window) After the Date of the Last Dose of Study Intervention or The First Date Starting a New Anticancer Therapy, whichever is Earlier

SECONDARY OUTCOMES:
Overall Survival | Time from randomization in a randomized Originator study, or from the first dose in a non-randomized Originator study, until death from any cause (Up to 93 Months)
  Overall survival is defined as the time from randomization in a randomized Originator study, or from the first dose in a non-randomized Originator study, until death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (36):
- United States (18):
  - Cancer Specialists, LLC, Jacksonville, Florida
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Florida Cancer Specialists, Sarasota, Florida
  - The Emory Clinic, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic- Minnesota, Rochester, Minnesota
  - University Of Nebraska Medical Center, Omaha, Nebraska
  - Cayuga Cancer Center, Ithaca, New York
  - Northwell Health, Lake Success, New York
  - Memorial Sloan-Kettering Cancer Center (MSKCC) - New York, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Tennessee Oncology, Nashville, Tennessee
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Swedish Cancer Institute, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (3):
  - Flinders Medical Centre, Adelaide
  - Peter MacCallum Cancer Centre, Melbourne
  - Linear Clinical Research, Victoria
- CHU de Nantes - Hotel Dieu, Nantes, France
- Italy (2):
  - IRCCS-AOU di Bologna-Policlinico S.Orsola-Malpighi, Bologna
  - Ospedale San Raffaele, Milan
- Japan (6):
  - Nagoya Medical Center, Aichi-Ken
  - National Cancer Center Hospital, Cho-ku
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Tokai University Hospital- Isehara Campus, Isehara
  - Tohoku University Hospital, Miyagi-Ken
  - Hokkaido University Hospital, Sapporo
- Poland (2):
  - Pratia MCM Krakow, Krakow
  - Instytut Hermatologii I Transfuzjologii, Warsaw
- Seoul National University Hospital, Seoul, South Korea
- United Kingdom (3):
  - St James's University Hospital, Leeds
  - Churchill Hospital, Oxford
  - Derriford Hospital, Plymouth

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/